CLINICAL TRIAL: NCT03597997
Title: Effects of Intraoperative Total Intravenous Anaesthesia (TIVA) With Propofol Versus Inhalational Anaesthesia on Postoperative Pain After Hepatectomy: a Randomized Controlled Trial
Brief Title: Effects of TIVA With Propofol Versus Inhalational Anaesthesia on Postoperative Pain After Hepatectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW18-176
Record Dates: First submitted 2018-06-28; First posted 2018-07-24 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Total intravenous anaesthesia; TIVA; Propofol; Hepatectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: Patients in one group (S) will be anaesthetized by inhalational anaesthesia using sevoflurane. The patients in the second group (P) will be anaesthetized using total intravenous propofol.
Who Masked: Participant, Investigator
Masking Description: Patients will not be aware of the type of anaesthesia they will receive. A separate blinded investigator will assess the patients after the operation. The anaesthetist providing general anaesthesia will be aware of the allocation, but s/he will not be involved in data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Experimental): The patients in group (P) will be anaesthetized using total intravenous propofol.
  Interventions: Drug: Propofol
- Group S (Sham Comparator): Patients in group (S) will be anaesthetized by inhalational anaesthesia using sevoflurane.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Target controlled infusion (TCI) with modified Marsh effect site model (Fresenius Kabi) will be used for induction and maintenance of general anaesthesia. Monitoring and other anaesthetic procedures including the management of hypertension and hypotension in group P will be the same as group S. The only difference is that induction and maintenance of general anaesthesia will be conducted using total intravenous infusion of propofol. Oxygen and air would be given to provide a FiO2 of 30-50%.
  Arms: Group P
Drug: Sevoflurane — Propofol 1.5-3mg/kg, remifentanil 1mcg/kg, and rocuronium 0.6-1mg/kg or atracurium 0.5mg/kg will be used intravenously for induction of general anaesthesia. Intubation would be performed after induction of general anaesthesia. General anaesthesia monitoring will be used. Sevoflurane, air and oxygen will be used for maintenance of general anaesthesia. FiO2 will be kept between 35-50%. BIS monitoring will be applied and level of anaesthetia will be titrated to maintain a BIS value of between 40-60. Intravenous remifentanil infusion between 0.1-0.2 mcg/kg/min will be given and this will be titrated to provide optimal haemodynamic parameters.
  Arms: Group S

SUMMARY:
Propofol is a commonly used intravenous anaesthetic drugs both for induction and maintenance of general anaesthesia. Advantages of total intravenous anaesthesia (TIVA) with propofol include reduced nausea and vomiting, reduced atmospheric pollution, and better wake up profile. But the need for a reliable intravenous access, specialized pumps, pain on injection and potential concerns regarding awareness are potential disadvantages of TIVA propofol.

Results from clinical trials have not been consistent. Some randomized trials have shown improved analgesia with TIVA propofol, and some reported no significant difference. A meta-analysis found that propofol was associated with a statistically significant reduction pain scores 24 hours after surgery. However, the clinical effect size was small. Therefore, the usefulness of propofol as an analgesic adjunct is still inconclusive.

Whether TIVA propofol is useful in providing significant postoperative analgesia may be influenced by the type of surgery and accompanying analgesic regime. This agrees with the concept of procedure specific analgesia. Liver surgery produces moderate to severe pain as a result of an upper abdominal incision. Pain control can be difficult due to concerns with epidural analgesia in patients with potential clotting abnormalities and the effect of analgesic metabolism as a in patients with liver dysfunction. Results from our retrospective study showed that TIVA propofol was associated with reduced pain scores with coughing on postoperative days 1 and 2, and also reduced opioid consumption when compared with sevoflurane after liver surgery.

In this study, the investigators plan to conduct a randomized controlled trial to further determine whether TIVA propofol reduces acute postoperative pain and opioid consumption after hepatectomy.

DETAILED DESCRIPTION:
* Preoperative care

Assessment will be done at the preadmission clinic or at the general ward. Fasting for patients will start at midnight before operation. Sedative premedication will not be prescribed.

* Anaesthesia and intraoperative care

= Group S (sevoflurane) - Patients from group S will be anaesthetized by inhalational anaesthesia using sevoflurane, according to the following protocol:

On arrival to the operation theatre, a 20 or 22 gauge intravenous cannula will be inserted. Standard monitoring with pulse oximeter, non-invasive blood pressure, and three lead electrocardiogram will be applied prior to induction. Non-invasive blood pressure will be checked at least every 5 minutes throughout the operation.

Propofol 1.5-3mg/kg, remifentanil 1mcg/kg, and rocuronium 0.6-1mg/kg or atracurium 0.5mg/kg will be used intravenously (IV) for induction of general anaesthesia. Intubation would be performed after induction of general anaesthesia. General anaesthesia monitoring will be used. Sevoflurane, air and oxygen will be used for maintenance of general anaesthesia. FiO2 will be kept between 35-50%. BIS monitoring will be applied and level of anaesthetia will be titrated to maintain a BIS value of between 40-60. Intravenous remifentanil infusion between 0.1-0.2 mcg/kg/min will be given and this will be titrated to provide optimal haemodynamic parameters. Muscle relaxants can be given during the operation as required.

Intravenous phenylephrine, ephedrine or fluid administration with colloid or crystalloid will be given at the discretion of the anaesthesiologist for management of hypotension. Hypertension or tachycardia will be managed by titrating the remifentanil infusion up to 0.2mcg/kg/min or sevoflurane up to 1.5 MAC. Intravenous anti hypertensive agents such as beta blockers (eg. esmolol, labetolol), hydralazine, glyceryl trinitrate, and phentolamine can be given if hypertension persists.

Thermal blanket will be used with the aim of keeping a core temperature of 35.5-37.5 degrees Celsius. Ondansetron 4mg IV will be given 30 minutes before end of surgery.

Sevoflurane and remifentanil infusion will be switched off at the end of the procedure. Reversal of muscle relaxation can be obtained if required with neostigmine 50mcg/kg IV and atropine 20mcg/kg IV after the operation. Patients will subsequently be transferred to the post anaesthetic care unit (PACU) for monitoring for at least 30 minutes.

= Group P (propofol) - Patients in group P will be anaesthetized using total intravenous propofol, according to the following protocol:

Monitoring and other anaesthetic procedures including the management of hypertension and hypotension will be the same as group S. The only difference is that induction and maintenance of general anaesthesia will be conducted using total intravenous infusion of propofol. Sevoflurane will not be used, and oxygen and air would be given to provide a FiO2 of 30-50%.

Target controlled infusion (TCI) with modified Marsh effect site model (Fresenius Kabi) will be used for induction and maintenance of general anaesthesia. Level of anaesthesia will be titrated to produce a BIS value of between 40-60. During induction of general anaesthesia, remifentanil 0.5-1mcg/kg, and rocuronium 0.6-1mg/kg or atracurium 0.5mg/kg will be given intravenously (IV). Remifentanil will be infused at a rate of between 0.1-0.2mcg/kg/min during maintenance of anaesthesia.

* Analgesic modalities and pain assessment

Both groups (Groups S and P)

Morphine sulphate at a bolus dose of 0.1mg/kg will be given intravenously before skin incision. Additional 0.1mg/kg of morphine sulphate can be given in divided doses when the surgery has continued for more than 2 hours at the discretion of the anaesthetist. Ketamine 0.5mg/kg intravenously will be given before skin incision. Patients will receive local wound infiltration with up to 2mg/kg of levobupivicaine during wound closure.

Resting pain scores will be checked every 5 minutes in the post anaesthetic care unit. 2mg boluses of intravenous morphine sulphate will be given every 5 minutes until the NRS pain score is less than 4/10. Respiratory rate, oxygen saturation, Ramsay sedation scores, blood pressure and heart rate will be monitored every 5 minutes while the patient is in the post anaesthetic care unit. A PCA morphine machine will be connected to the patient once the NRS pain score is less than 4/10. The PCA morphine machine will be set to give 1mg of intravenous morphine sulphate with each patient demand, and lockout duration of 5 minutes will be set. Maximum dose limit will be 0.1mg/kg of morphine sulphate per hour and basal infusion will not be given.

When the patient resumes fluid diet in the ward on postoperative day 0, regular oral dihydrocodeine will be prescribed at a dose of 30mg tds for two days. Afterwards, dihydrocodeine will be given as needed. Breakthrough pain will be treated by intramuscular/subcutaneous morphine 0.1mg/kg every 4 hours as needed starting from postoperative day 0.

Respiratory rate, oxygen saturation, sedation scores will be monitored every hour while patient is using PCA morphine. Blood pressure and heart rate will be measured every 4 hours. Pain related parameters like the numerical rating scales (NRS) pain scores at rest and during cough, cumulative PCA morphine doses and number of PCA demands/goods delivered, and side effects will also be recorded very 4 hours. Anaesthesiologists will assess patients every day to determine the adequacy of analgesia.

PCA morphine will be given for at least 2 days. PCA morphine will be stopped on postoperative day 2 if NRS pain scores during cough is less than 4/10 and morphine consumption is low. If PCA morphine consumption is high or NRS pain scores during cough is equal or greater than 4, PCA morphine will be continued. Assessment will be performed everyday. An NRS pain score that is 4 or higher during coughing on postoperative day 5 will require an evaluation for complications. The patient will be further managed at the discretion of the anaesthesiologist. After discontinuation of PCA morphine, NRS pain scores (at rest and with coughing) and the dose and frequency of rescue analgesia used will be recorded daily until patient discharge.

NRS pain score and satisfaction with analgesia (scored from 0-10, where 0 is the least satisfaction and 10 most satisfaction) will be obtained.

Quality of recovery 9 (QoR-9) is measured at 24h and 72h after surgery. The attending surgeon will determine final hospital discharge

* A brief home telephone interview will be conducted at 3 and 6 months to assess the incidence of chronic pain. The severity of pain, if present, would be recorded using NRS (0-10) at rest and with coughing. Other information that will be obtained at 3 and 6 months after surgery include HRQOL obtained with the Chinese-HK version of the SF12v2- health survey and psychological condition will be assessed with the Hospital Anxiety and Depression Scale (HADS) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* ASA I to III
* Scheduled for elective hepatectomy (left or right hepatectomy, segmentectomy, or wedge resection)

Exclusion Criteria:

* Known drug allergy to propofol, opioids, non-steroidal anti-inflammatory drugs (NSAIDs) including COX-2 inhibitors, paracetamol, ketamine
* Alcohol or drug abuse
* Impaired renal function, defined as preoperative serum creatinine level over 120µmol/L
* Impaired or retarded mental state
* BMI > 35kg/m2
* History of chronic pain
* Pregnancy
* Local infection
* History of psychosis, delirium
* Chronic opioid user
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Pain assessed by numercial rating scales (NRS) pain scores | at postoperative day 1
  NRS pain scores (from 0-10, where 0 is the least satisfaction and 10 most satisfaction) will be recorded at rest and with coughing everyday.

SECONDARY OUTCOMES:
PCA morphin consumption | from postoperative day 0 until postoperative day 5
  Cumulative PCA morphine doses (in mg) will be recorded daily based on medical record.
Dihydrocodeine use | from postoperative day 0 until postoperative day 5
  Frequency of dihydrocodeine use (i.e. how many times per day) will be recorded daily according to medical record.
Side effects of analgesics | from postoperative day 0 until postoperative day 5
  Pruritus, dizziness, nausea, vomiting, wound infection, urinary retention, confusion, constipation will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Stanley SC Wong, MBBS, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wong SSC, Wang F, Chan TCW, Cheung CW. The analgesic effect of total intravenous anaesthesia with propofol versus inhalational anaesthesia for acute postoperative pain after hepatectomy: a randomized controlled trial. BMC Anesthesiol. 2023 Apr 3;23(1):112. doi: 10.1186/s12871-023-02063-7. PMID 37013472